CLINICAL TRIAL: NCT04180085
Title: Pilot Study: Interest of Belatacept as a Non-nephrotoxic Immunosuppressive Treatment in Cardiac Transplant Patients at Risk of Chronic Renal Failure
Brief Title: Pilot Study: Interest of Belatacept as a Non-nephrotoxic Immunosuppressive Treatment in Cardiac Transplant Patients at Risk of Chronic Renal Failure (BELACOEUR)
Acronym: BELACOEUR
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC19_0133
Record Dates: First submitted 2019-11-25; First posted 2019-11-27 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Heart Transplant Failure
MeSH Terms: interventions — Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BELATACEPT (Experimental)
  Interventions: Drug: Belatacept Injection

INTERVENTIONS:
Drug: Belatacept Injection — 9 injections of belatacept at 3 months, 4 months, 5 months, 6 months, 7 months, 8 months, 9 months, 10 months 11 months and 12 months post graft

SUMMARY:
Heart transplantation (TC) is the standard treatment for terminal heart failure. Chronic kidney disease (CKD) is a common complication responsible for increased mortality and morbidity. The main risk factors for progression to CKD are advanced age, pre-transplantation CKD, degradation of glomerular filtration rate (GFR) in the first year post-transplantation, and nephrotoxicity of calcineurin inhibitors (CNI).

Indeed, these molecules (cyclosporin and tacrolimus), the cornerstone of immunosuppressive treatment, have nephrotoxic effects in the short term (by a hemodynamic effect) and in the long term (by a pro-fibrosin effect).

In renal transplantation (TR), belatacept, a costimulation-inhibiting molecule, used de novo, without CNI, with induction by anti-receptor antibody of Interleukines 2, preserves kidney function. Despite this great advantage, its development is still hampered by a higher number of rejections compared to the CNI group in this originator study. Based on the experience gained in TR, which has since validated its use, the hypothesis is that in heart transplantation, belatacept (Nulojix) combined with minimization of CNI (with induction by antilymphocyte serum), could significantly improve glomerular filtration rate (GFR) in patients at risk of CKD (by removing them from dialysis and possible kidney transplantation) without increasing the risk of rejection.

ELIGIBILITY:
Inclusion Criteria:

Cardiac transplant patients for 3 months Over 18 years of age No Donor Specific Antibodies at inclusion (positive threshold average fluorescence intensity (MFI)> 2000) Having a GFR (DFG in french) is the single best indicator of overall renal function < 30ml/min calculated according to the formula CKD EPI or a decrease in GFR of more than 50% between the day of the heart transplant and 3 months, stable for 15 days.

Induction treatment with anti-lymphocyte serum Virus d'Epstein-Barr positive serology Having signed the consent after receiving informed information Negative pregnancy test for patients of childbearing age, and agreement to use effective contraception throughout the study and 6 weeks after the end of the study Having no difficulty in understanding and communicating with the investigator and his representatives Beneficiaries of a Social Security scheme

Exclusion Criteria:

The criteria for non-inclusion are:

2nd heart transplant or other solid organ transplant History of rejections Cellular or humoral rejection at myocardial biopsy of 3 months post Transplantation Cardiac Current viral infection of type cytomegalovirus, Virus d'Epstein-Barr, hepatitis C virus, hepatitis V virus.....

Human immunodeficiency virus positive serology Ongoing participation in another clinical study Any clinical condition that the investigator considers incompatible with the conduct of the study under acceptable safety conditions: (in particular, progressive infection, progressive cardiovascular complication, progressive neoplastic disease) Inability of the patient to comply with study procedures Pregnant or breastfeeding women Person under guardianship, curators or safeguard of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-02-06 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Clearance | 12 months
  Determination of plasma creatinine and calculation of clearance according to the formula CKD EPI (Chronic Kidney Disease - Epidemiology Collaboration) at 3 months and 12 months post heart transplantation

SECONDARY OUTCOMES:
Myocardial biopsies | 12 months
  Myocardial biopsies between 3 months and 12 months post Cardiac Transplantation to check the risk of rejection
Anti-human leukocyte antigen antibody assay | 12 months
  To check the risk of rejection
Fasting blood glucose and glycated haemoglobin (HBA1C) | 12 months
  Measurement of the New Onset Diabetes After Transplantation
Death | 12 months
  Evaluate the mortality specific to 12 months post cardiac transplantation (Estimate: percentage of patients who died at 12 months).
Number of dialysis sessions | 12 months
  Evaluate the use of renal replacement therapy between 3 months and 12 months after Cardiac Transplantation.

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Karine Nubret, Bordeaux
  - Laurent Sebbag, Lyon
  - Claire Garandeau, Nantes
  - Bertrand Lelong, Rennes